CLINICAL TRIAL: NCT01104181
Title: Collection of Anal Specimens for Assessment of Anal Cancer Using the HC2 High-Risk DNA Test (QIAGEN)
Brief Title: Hybrid Capture 2 Human Papiloma Virus (HPV) High-Risk Anal DNA Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laser Surgery Care (Other)
Collaborators: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Stephen E. Goldstone, M.D., Laser Surgery Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: R09-HPV-001
Record Dates: First submitted 2010-03-25; First posted 2010-04-15 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Anal Canal HPV Infection Diagnosis; Anal Dysplasia Diagnosis; Anal Cancer
Keywords: Anal HPV; Anal Dysplasia; Ana Cancer
MeSH Terms: conditions — Anus Neoplasms | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- swab and brush or swab and swab (Experimental): we will determine which collection method is superior
  Interventions: Device: HC2 collection kit with a swab or brush

INTERVENTIONS:
Device: HC2 collection kit with a swab or brush — We will sample the anal canal for cells with either a swab and swab or swab and brush to determine which is superior
  Other Names: Qiagen HC2 HPV High-Risk DNA Test

SUMMARY:
This is a study to determine if HC2 HPV testing in the anal canal can detect high-risk HPV and whether this aids in identifying individuals are risk for anal cancer or precancerous lesions.

ELIGIBILITY:
Inclusion Criteria:

1. male or female 18 years of age or older
2. screened for anal dysplasia, including MSM and women -

Exclusion Criteria:

1. subject has had a previous treatment for anal cancer.
2. subjects that have used enemas or other foreign substances, in the anal canal or anal sex within 24 hours of collection.
3. subjects that have bleeding disorders or use anticoagulation treatments. -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
HC2 can accurately test for oncogenic HPV in anal specimens | in approximately 12 months
  Determination that HC2 testing in the anal canal can be performed

SECONDARY OUTCOMES:
Sensitivity and specificity of cytology with HC2 | in approximately 12 months
  To determine if HC2 improves the sensitivity and specificity of anal cytology

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Goldstone, MD, Principal Investigator — Mount Sinai Medical School
Locations (1):
- Laser Surgery Care, Inc., New York, New York, United States